CLINICAL TRIAL: NCT06183905
Title: A Prospective Cohort Study Comparing Multi-parametric Ultrasound Versus Multi-parametric MRI for Clinically Significant Prostate Cancer Detection
Brief Title: Multi-parametric Ultrasound Versus Multi-parametric MRI for Prostate Cancer Detection
Acronym: TRUSVSMPMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XH-23-012; 21y11911000 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality)
Record Dates: First submitted 2023-11-23; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-11

CONDITIONS: PROSTATE CANCER; Prostate Biopsy
Keywords: prostate cancer; multiparametric ultrasound; multiparametric MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging (multiparametric ultrasound and multiparametric MRI) (Experimental): All patients will undergo multiparametric ultrasound and multiparametric MRI. In case of suspicious multiparametric ultrasound and/or multiparametric MRI,they will undergo combined targeted biopsy and systematic biopsy. In case of nonsuspicious imaging findings, only systematic biopsy will be performed.
  Interventions: Diagnostic Test: Prostate imaging; Procedure: Prostate biopsy

INTERVENTIONS:
Diagnostic Test: Prostate imaging — Multiparametric ultrasound (mpUS) The mpUS examinations are performed in the order of greyscale imaging, elastography and contrast-enhanced ultrasound (CEUS), with the patients in the left lateral decubitus position.Greyscale imaging and elastography are evaluated by one radiologist. After standard step-sectional greyscale imaging, transverse elastic images are obtained from the base to the apex by manual compression. The amplitude and frequency of compression are adjusted according to the visual compression indicator on the screen to minimize interoperator variability. CEUS is performed using a bolus of 2.4 mL contrast agents (SonoVue, Bracco) using Contrast mode.
  Multiparametric MRI (mpMRI) Prostate mpMRI images were acquired using a 3-T scanner with an external phased-array coil.
Procedure: Prostate biopsy — All patients will undergo standard 12-core systematic biopsy (SB) within 1 week following the imaging protocol in conjunction with targeted biopsy (TB) for suspicious lesions on mpUS and/or mpMRI. First, 12-core SB is performed, followed by cognitive mpUS-TB with 2-3 cores for each suspicious lesion. The suspicious lesions on mpUS include hypoechoic lesion(s) on greyscale imaging, reproducible stiff lesion(s) on elastography, and hypoperfused area(s) with ill-defined boundaries or increased focal/asymmetric contrast enhancement on CEUS. Thereafter, MRI/US fusion TB is performed sampling 2-3 cores for each lesion with a Prostate Imaging Reporting and Data System (PI-RADS) version 2 score of 3 or above.Each biopsy sample is placed in the micro-cassette and labelled to identify the biopsy technique and location.

SUMMARY:
The goal of this cohort study is to investigate multiparametric ultrasound versus multiparametric MRI for clinically significant prostate cancer detection in patients scheduled for initial biopsy. The main questions it aims to answer are:

* whether the clinically significant prostate cancer detection rate of multiparametric ultrasound is comparable to multiparametric MRI
* the any cancer detection of multiparametric ultrasound versus multiparametric MRI

Participants will undergo multiparametric ultrasound and multiparametric MRI before prostate biopsy. In case of suspicious findings on ultrasound or MRI, they will undergo combined systematic biopsy and targeted biopsy. In case of nonsuspicious imaging finding, they will undergo systematic biopsy alone.

DETAILED DESCRIPTION:
In recent years, the multi-parametric MRI targeted biopsy showed inspiring results for improving clinically significant prostate cancer (PCa) detection rate [1]. Two techniques have been developed for MRI targeted prostate biopsy: in-bore MRI guided biopsy and MRI/ultrasound fusion biopsy. However, these biopsy techniques require specific equipment and software. Moreover, MRI has contradictions and cannot be performed in all patients. Therefore, an imaging targeted biopsy adjunct to MRI targeted biopsy is needed.

Besides MRI, multi-parametric ultrasound can also visualize PCa lesions by providing information about the blood supply, perfusion and stiffness of the prostate gland for PCa detection. Our hypothesis is as follows, (1) clinically significant PCa detection rate by multi-parametric ultrasound targeted biopsy is comparable with multi-parametric MRI targeted biopsy; (2) clinically significant PCa detection rate by either multi-parametric ultrasound targeted biopsy or multi-parametric ultrasound targeted biopsy is higher than standard systematic biopsy. Our secondary outcome also includes the any cancer detection rate and clinically insignificant prostate cancer detection rate.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for prostate biopsy;
2. Signed the informed consent.

Exclusion Criteria:

1. Contraindications to MRI, such as metal implants, claustrophobia, etc;
2. Contraindications to ultrasound, such as acute myocardial infarction, acute cerebral infarction and rectal tumor after Miles operation;
3. Contraindications of prostate biopsy, such as abnormal routine urine test, coagulation function and electrocardiogram
4. Any medical condition or other event that may significantly reduce the chances of obtaining reliable data, achieving the purpose of the study or completing the study and follow-up;
5. The study doctor thinks it is not suitable to participate in this study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
clinically significant prostate cancer detection | Up to 12 weeks following imaging
  The primary definition was Grade Group(GG) ≥ 2. The secondary definition included PROMIS definition 1 (GG ≥ 3 and/or maximal cancer core length ≥ 6 mm) and PROMIS definition 2 (GG ≥ 2 and/or maximal cancer core length ≥ 4 mm). The measurement that will be based on biopsy histopathology.

SECONDARY OUTCOMES:
Any cancer detection | Up to 12 weeks following imaging
  Any cancer at biopsy histopathology. The measurement that will be based on biopsy histopathology.
Clinically insignificant prostate cancer detection | Up to 12 weeks following imaging
  Clinically insignificant prostate cancer at biopsy histopathology. The measurement that will be based on biopsy histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Yunkai Zhu, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
individual participant data are only available from the investigator on reasonable request